CLINICAL TRIAL: NCT05372497
Title: Effect of Central Nervous System Focused Therapy in Frozen Shoulder Patients: A Randomized Controlled Trial
Brief Title: Central Nervous System Focused Therapy in Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, AYŞE GÜRLÜK, Physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedipolUniversity2020
Record Dates: First submitted 2022-04-27; First posted 2022-05-12 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2023-12

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physiotherapy plus central nervous system focused treatment group (CP+CNS group) (Experimental): For the patients participating in the study, a protocol focused on the central nervous system and aimed at reducing hypersensitivity was applied with pain, graded sensory discrimination and graded motor imagery (GMI) training in addition to conventional physiotherapy. Graded sensory dicrimination training includes localization training level 1, localization training level 2 and graphesthesia training. GMI training includes right/left discrimination training, visual imagery, isometric and functional exercises, and mirror therapy. The treatment was applied in 20 sessions, for 45-60 minutes, 5 days a week.
  Interventions: Other: Intervention group (IG)
- Conventional Physiotherapy Group (CP Group) (Active Comparator): In the conventional physiotherapy group of the study, in addition to physiotherapy modalities for 20 sessions, 5 days a week, for 45-60 minutes each session, 5 days a week, electrotherapy, scapular mobilization, passive stretching, stick exercises, finger ladder exercises, pendulum exercises and shoulder flexion, extension, abduction, internal rotation, external rotation strengthening exercises were applied.
  Interventions: Other: Control group (CG)

INTERVENTIONS:
Other: Intervention group (IG) — Participants randomized to this treatment will receive a central nervous system-focused intervention consisting of a 20-session treatment program delivered in 30-45-minute sessions scheduled 5 days a week over a 4-week period and standard physical therapy will be continued.
  * Chronic pain training will be given according to the needs of the person and 5-10 minutes will be allocated every day for the first week and chronic pain education will be divided into modules.
  * Right / Left Discrimination Training
  * Localization Training Level 1- Level 2 Training
  * Visual imagination Training
  * Visual Imagery Training
  * Mirror Therapy
  * Isometric and functional exercises
  Arms: Conventional physiotherapy plus central nervous system focused treatment group (CP+CNS group)
Other: Control group (CG) — The control group will receive only conventional physiotherapy. Conventional physiotherapy will be 5 days a week.
  The conventional physiotherapy treatment session will take place as follows.
  * Electrotherapy
  * Scapular mobilization
  * Passive stretches
  * Stick Exercises
  * Pendulum Exercises
  * Shoulder flexion, extension, internal rotation, external rotation, horizontal abduction/ adduction strengthening exercises
  Conventional physiotherapy intervention is planned for 45-60 minutes a day, five days a week for both groups.
  Arms: Conventional Physiotherapy Group (CP Group)

SUMMARY:
Frozen shoulder has been considered a self-limiting and benign disease with complete resolution of pain and ROM, but this can sometimes last for years. This prolonged pain and disability deprives patients of their routine life, occupational and recreational activities. Although appropriate treatment is needed so that they can quickly return to their lives, definitive treatment strategies have not been established and many different management strategies are used. The aim of this study is to investigate whether pain education and sensory education applied together with conventional physiotherapy are more effective than conventional physiotherapy alone.In this study, 21 people diagnosed with frozen shoulder who were referred by the doctor of Esenler Medipol Hospital, Department of Physical Therapy and Rehabilitation will be included in the study.

Outcome measures: Pain Beliefs Scale, Pain Catastrophizing Scale, PainDetect Questionnaire, Tampa Kinesiophobia Scale, Shoulder Pain and Disability Index, Visual Analog Scale, Electrogoniometer, Two-point discrimination test, Numeric Rating Sleep Scale and Right/ Left Judgement Task.

This study was designed as a prospective randomized controlled trial. 21 people were included in the study. Participants were randomly divided into two groups: Conventional physiotherapy group (CP group) (n=11), Conventional physiotherapy plus central nervous system focused treatment group (CP+CNS group) (n=10). Conventional physiotherapy was applied to both groups for 45-60 minutes, 5 days a week for 4 weeks.

The CP group treatment session will take place as follows: Scapular mobilization, passive stretches, stick exercises, pendulum exercises and shoulder flexion, extension, internal rotation, external rotation, horizontal abduction/ adduction strengthening exercises.

The CP+CNS group received central nervous system focused therapy that included chronic pain education, localization training, graphesthesia, graded motor imagery and mirror therapy in addition to conventional physiotherapy.

The IG group protocol includes:

1. week: Initial Evaluation, Conventional physiotherapy (CP), Chronic Pain Education, Localization Training Level 1, Right / Left Discrimination Training
2. week: CP, Motor Imagery, Localization Training Level 2
3. week: CP, Grafestesis Training, Isometric Exercise
4. week: CP, Mirror Therapy, Functional Exercises, Final Evaluation

DETAILED DESCRIPTION:
First week:

* Initial Evaluation
* Conventional physiotherapy (CP) (5 days)
* Chronic Pain Education (5 days):Chronic pain education is a therapeutic treatment strategy that explains the patient's past experiences of pain in terms of neurobiological and neurophysiological rather than anatomical or biomechanical models. Detailed chronic pain education is needed to redefine the concept of pain and to convince the patient that the cause of their symptoms is hypersensitivity of the central nervous system rather than local tissue damage. For this reason, chronic pain education modules were created by the researcher to be presented to the participants in order to change their pain beliefs through the reconceptualization of pain. Nociceptive mechanisms in acute pain and chronic pain were explained comparatively at the beginning. A presentation supported by visuals and examples was prepared to guide during the chronic pain education, but a flexible schedule of 15-20 minutes was created by increasing the number of examples and in more detail according to the education level of the patient, preventing the patient from being bored during the session.
* Localization Therapy Level 1 (5 days): This level only the localization of the stimulus was trained. A grid-like sticky paper with 9 holes punched was placed over the affected shoulders of the participants and the training began by showing a standard photograph of the shoulder on which the 9-hole grid was marked. The spacing of the grids was determined on the basis of available data based on two-point separation of the shoulder joint.This data range was 43.18 mm ± 10.37 mm. The standard limits for placement of the 9-hole grid on the shoulder are as follows: 1 cm proximal to the acromioclavicular joint and the lower border of the insertion of the deltoid muscle. The thick end of the probe and the 9-hole grill and their placement on the shoulder are introduced. After the familiarization period, the patient continues training with the thick end of the probe (2 seconds) using a random number sequence. In the first week, stimulus was applied by asking random numbers 4 days a week, 3 sets every day and 20 numbers in each set.
* Right / Left Discrimination Training (5 days): In the first week, an online computer program, Recognise Shoulder (Recognise Online, NOI Group, Adelaide, SA, Australia) was used to present participants with randomly selected photographs of their right or left shoulder. Shoulder photos presented in various directions. Participants were asked to press one of the buttons on the left and right of the screen to indicate whether the photograph was of the right or left shoulder. An important point here was to give the response corresponding to the body part as quickly as possible, and for this purpose, the participants were asked to respond within 5 seconds during the application. The training was carried out in three sets, each set consisting of 30 photographs.

Second week:

* Conventional physiotherapy (CP)
* Motor Imagery (5 days): In our study, participants were asked to imagine they were moving their painful shoulders with motor imagery training. Participants were asked to sit in a comfortable position, close their eyes, and imagine being in an environment where they felt comfortable. Photographs containing 8 shoulder postures were used in the training. 8 photos were applied in two sets and 20 repetitions. Each photograph was shown live to the participants by the physiotherapist and the participant was asked to imagine the motion shown as painless, smooth and full range of motion. Participants were asked not to imagine watching themselves while imagining shoulder movements, but to perform the movements in the first person.
* Localization Training level 2 (5 days): They were asked to distinguish both the localization of the stimulus and the size of the probe used. The working pattern is the same as for localization level 1, but two types of probes are used, pointed (pencil tip) and coarse tip (mushroom). Three randomly applied sets of both position and probe sizes and a random array of 20 numbers in each set were used.

Third week:

* Conventional physiotherapy
* Grafestesis Training (5 days): In our study, randomized capital letters were drawn consecutively on the affected shoulder of the participant by the physiotherapist using the index finger. On the second day, the randomized letters were drawn in lowercase and the patient was asked to say the correct letter. On the third day, the randomized letters drawn on the shoulder were presented in different directions and the participant was asked to say the correct letter. On the fourth day, random letters were presented in slow, fast, and normal speed and the participant was asked to say the correct letter. On the fifth day, 20 meaningful words consisting of three letters were formed. It was written overlapping the participant's shoulder and the patient was asked to say the meaningful word.
* Isometric exercise (5 days): Three sets of isometric exercises including shoulder flexion, extension, abduction and adduction movements, each set consisting of 7-10 repetitions and each movement lasted for 10 seconds, were performed. The participant completed the movements with controlled breathing while performing the movements, and a 1-3 minute rest break was given between each set.

Fourth week:

* Conventional physiotherapy
* Mirror Therapy (5 day): A large mirror with wheels was placed in front of the participant with the unaffected arm facing the reflective side of the mirror, and the participant was allowed to flex the trunk to see the unaffected arm. Mirror therapy initially began with the unaffected arm watching its movements on the moon. It was said that when the participant was confident that he could do the mirror exercises painlessly, he could start performing the movements with the affected shoulder at the same time. Afterwards, progress was made towards active movements involving shoulder flexion, abduction, internal rotation and external rotation, including the affected arm. In the clinic, a training was planned for 2 sets, lasting 12-15 minutes, and rest periods of 1-3 minutes between each set.
* Functional Exercises (5 day): The movements that the participant had difficulty in daily life were determined during the individual interview, and exercises similar to these movements and specifically aimed at increasing functionality were planned in the clinic and applied for 15 minutes. Functional exercises wiping the wall opposite the wall at different degrees of flexion and abduction in close and far distances, wiping the wall with narrow and wide circumcision movements, picking up colored papers placed on the mirror at different angles and placing them at different angles, squeezing the ball while shoulder flexion and abduction involved rolling the ball wide and narrow with the shoulder at different angles.
* Final Evaluation

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with frozen shoulder with chronic pain lasting more than 3 months
* Being between the ages of 18-65
* Absence of fracture, dislocation or arthritis in the shoulder area evaluated by routine x-ray examination
* Patients who were not prescribed any medical treatment other than analgesics in the last 3 months were included.

Exclusion Criteria:

* Wide scar around the shoulder
* History of bilateral concurrent frozen shoulder
* If there has been surgical intervention on the affected shoulder
* Rotator cuff calcification
* Cervical radiculopathy
* History of physical therapy program for the same shoulder in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
The Pain Catastrophizing Scale | Change from The Pain Catastrophizing Scale at 4 weeks
  The PCS is used to evaluate the patient's feelings, thoughts, and emotions related to pain and catastrophizing. it is a self-administered questionnaire with 13 items and 3 subscales: helplessness, magnification, and rumination. A 5-point scale is used for each item, with higher values representing greater catastrophizing. The scores for each item are added to determine the subscales, and the total score is calculated by the summation of all items. The PCS scores range from 0 to 52 points
Visual Analog Scale (VAS) | Change from Visual Analog Scale (VAS) at 4 weeks
  It is used to assess pain. Although pain has been defined in many different ways, the most widely accepted is the International Association for the Study of Pain (IASP); It is a definition of "sensory, emotional, unpleasant feeling related to the past experiences of the person, whether due to an organic cause originating from any part of the body or not" (20). Visual Analogue Scale (VAS) is a reliable and valid pain measurement method in the evaluation of the severity of chronic pain (21). There is a numeric horizontal line between zero and ten. Zero means "no pain" and ten means "unbearable pain". Below the horizontal scale are facial expressions.
Electrogoniometer | Change from electrogoniometer at 4 weeks
  Normal joint movements measurement is evaluated with active or passive movements. The most used instrument for the objective evaluation of these movements is the electrogoniometer. All joints are placed according to the anatomical position before measurement and this position is considered as the zero initial position. The electrogoniometer should not touch the body during measurement and should be placed lateral to the joint. In this study, shoulder joint electrogoniometer measurements will be made. Shoulder flexion, abduction, internal rotation, external rotation will be measured at the beginning and at the end of the 4th week, with an electrogoniometer, normal range of motion will be measured.
Two Point Discrimination Test | Change from two point discrimination test at 4 weeks
  The two-point discrimination test is the evaluation of the ability to perceive stimuli applied from two different points at the same time. A commercially available mechanical caliper will be used to measure two-point separation on the non-dominant and dominant shoulders. These areas within the shoulder will correspond to the C5, C6 and C7 dermatomes. Participants will be instructed to report to the tester if they repeatedly feel two points or if the pressure is greater than a light touch.Care should be taken that the warning given while performing the test does not cause pain. Evaluation will be made with the aid of an esthesiometer. The esthesiometer is used to measure the person's 2-point sensory threshold on the skin. The ruler opens until you feel the 2 points and the value is recorded.
Pain Beliefs Scale | Change from pain beliefs scale at 4 weeks
  It was developed by Edwards et al. in 1992. They mention that the most important purpose of developing the scale is to understand the psychological and organic attributions of chronic pain patients to the origin of pain, which have not been investigated until that time. In the original form of this scale, there are a total of 20 items covering beliefs about the sources of pain and the treatment method. Two subtests were created: Organic Beliefs subtest consisting of 8 items and Psychological Beliefs subtest consisting of 4 items.
  Scores range from 1 to 6 for each item. The total score for each subtest is calculated by adding the scores obtained from the items in that subtest and dividing by the number of items belonging to that subtest.
Right/left Judgement Task | Change from right/left judgement task at 4 weeks
  For laterality assessment, SSDG was assessed with the Neuro Orthopedic Institute (NOI) Recognise Shoulder™ online program using an iPad. In order to gain familiarity, individuals were asked to mark whether 15 photos from the rapid test category belonged to the right or left shoulder. In the actual assessment, they were asked to answer 30 shoulder photos from the rapid test category as right and left as soon as possible. Mean response times (RT) in milliseconds (ms) and percentage of correct responses were reported separately for both the affected and unaffected shoulder region as the two main outcome measures. Responses below 500 ms and above 15000 ms were considered invalid.

SECONDARY OUTCOMES:
Tampa Kinesiophobia Scale (TKS) | Change from tampa kinesiophobia scale (TKS) at 4 weeks
  The Tampa Kinesiophobia Scale (TKS) was originally developed by Miller, Kopri, and Todd in 1991 but was not published. Vlaeyen et al. republished the original 17-question scale in 1995 with permission from the researchers who developed it. The validity and reliability study of the Turkish version was conducted by Yılmaz et al. in 2011. TKS is a 17-item scale developed to measure fear of movement/re-injury. The scale includes parameters of injury/re-injury and fear-avoidance in work-related activities. A 4-point Likert scoring (1=I totally disagree, 4=I totally agree) is used in the scale. After reversing the 4th, 8th, 12th and 16th items, the total score is calculated. The person gets a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia.
Shoulder Pain and Disability Index (SPADI) | Change from shoulder pain and disability index (SPADI) at 4 weeks
  The functional status of the patients was evaluated using the "Shoulder Pain and Disability Index". Shoulder pain and disability index is a questionnaire developed to measure shoulder pain-related pain and disability, consisting of two parts, pain and disability, and containing a total of 13 questions. There are 5 questions in the subgroup of the questionnaire that evaluates pain, and the patient is asked to express the severity of his pain during different activities in the last week by scoring between zero (no pain) and 10 (the most severe pain). In the subgroup in which disability is evaluated, there are 8 questions and the patient is asked to rate how much difficulty he has had during the different activities he has done in the last week, between zero (no difficulty) and 10 (receiving help). A total score of zero indicates maximum well-being, and 130 points indicate maximum ill health.
Pain Detect (PD-Q) | Change from shoulder pain detect (PD-Q)at 4 weeks
  The PD-Q is a simple questionnaire that allows the detection of neuropathic pain components in patients with chronic pain. PD-Q consists of four main parts. In the first part, it evaluates the intensity of current pain, the average and maximum pain intensity over the past 4 weeks. In the second part, patients are asked to mark one of the four graphs that best describe their pain course patterns. The third section includes a sensory map representing the homunculus, a bidirectional item about the presence of radiating pain, and questions that attempt to mark the area of pain with an arrow pointing in the direction of the radiating pain. In the last part, there are seven Likert-type items asking the intensity of the sensation marked on the homunculus. This last section provides scores between 0 and 35 points. The final score is obtained by adding the total scores of the last three sections from -1 to 38. PD-Q uses two cut-off values.
Graded Chronic Pain Scale-Revised | Change from graded chronic pain scale-revised at 4 weeks
  Persons with chronic pain are placed at grades 1, 2, or 3. Among persons with chronic pain, those who report that pain limits their life activities or work on most days or every day in the past 3 months (item 2) are placed at grade 3 (high-impact chronic pain). Among the remaining persons with chronic pain, those with a PEG total score of 12 or greater are placed at grade 2 (bothersome chronic pain). Those with chronic pain that is not high impact and whose PEG score is less than 12 are placed at grade 1 (mild chronic pain).
Sleep Scale | Change from sleep scale at 4 weeks
  A scale of zero to ten points will be used to assess sleep quality. The person will be asked to score between 0-10 points for sleep quality, considering how many hours they sleep, how easily they fall asleep, how often they wake up at night (except to go to the bathroom), how often they wake up early in the morning without having to, and how refreshing their sleep is. 0 means "terrible", 1-2-3 means "poor", 4-5-6 means "balanced", 7-8-9 means "good", 10 means "great".

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe GÜRLÜK, MSc, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University Esenler Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No